CLINICAL TRIAL: NCT06742736
Title: EXACERBATIONS AND REAL-WORLD OUTOMES INCLUDING CARDIOPULMONARY EVENTS AMONG PATIENTS WITH CHRONIC OBSTRUCTIVE PULMONARY DISEASE INITIATING BUDESONIDE/GLYCOPYRRONIUM/FORMOTEROL (MITOS: EROS+CP US Study)
Brief Title: EXACERBATIONS AND REAL-WORLD OUTOMES INCLUDING CARDIOPULMONARY EVENTS AMONG PATIENTS WITH CHRONIC OBSTRUCTIVE PULMONARY DISEASE (MITOS: EROS+CP US Study)
Acronym: EROS+CP (US)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00095
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Retrospective; Real-World Effectiveness
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Prompt: PATIENTS INITIATING BGF WITHIN 30-DAYS OF EXACERBATION
  Interventions: Drug: BGF
- DELAYED: PATIENTS INITIATING BGF WITHIN 31-180 DAYS OF EXACERBATION
  Interventions: Drug: BGF
- VERY DELAYED: PATIENTS INITIATING BGF WITHIN 181-365 DAYS OF EXACERBATION
  Interventions: Drug: BGF

INTERVENTIONS:
Drug: BGF — BUDESONIDE/GLYCOPYRRONIUM/FORMOTEROL
  Other Names: BREZTRI

SUMMARY:
A retrospective real-world data study, assessing the relationship between the timing of Budesonide/Glycopyrrolate/Formoterol initiation following an exacerbation and the occurrence of subsequent exacerbations, severe cardiopulmonary events and other real-world outcomes in the United States

ELIGIBILITY:
Inclusion Criteria:

* 1 prescription(s) fill for BGF on or following July 24, 2020 (date of BGF approval in the United States)

  * Patients must have evidence a qualifying exacerbation events which, per local or global guidelines, would qualify a patient to have treatment escalated or initiated to triple therapy. The qualifying exacerbation event must occur within the 12-month period preceding the initiation of BGF but occurring on or following local BGF commercial availability (July 24, 2020) and includes either of the following
* 12 months of continuous health plan enrollment preceding the qualifying index exacerbation event date ('baseline' period)
* 1 day of continuous enrollment following the qualifying index exacerbation date

  * Age ≥ 40 years on the qualifying index exacerbation event

Exclusion Criteria:

* Presence of cancer diagnoses other than basal or squamous cell skin cancer during the baseline or follow-up periods
* Presence of interstitial fibrosis, sarcoidosis, or pulmonary embolism diagnoses during the baseline or follow-up periods
* Presence of triple therapy SITT during the baseline period through BGF initiation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The overall sample will include adult (aged 40+) COPD patients who have experienced a qualifying COPD exacerbation and eventually received treatment with BGF. Patients should not have prior single inhaler triple therapy (SITT) use during the 12-month period-baseline prior to the qualifying index exacerbation and prior to initiating BGF treatment.
Sampling Method: Non-Probability Sample
Enrollment: 13000 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Annualized COPD Exacerbation Event Rate | Annualized rates from index exacerbation through end of data availability, mean follow-up 462 days
  Annualized rates of COPD exacerbation events observed from index date (qualifying exacerbation event) through study completion (or until end of data availability; mean follow-up 462 days

SECONDARY OUTCOMES:
Annualized Cardiopulmonary Event Rate | Annualized rates from index exacerbation through end of data availability; mean follow-up 462 days
  Annualized rates of cardiopulmonary events observed from index date (qualifying exacerbation event) through study completion (until end of data availability)

OTHER OUTCOMES:
Annualized rate of all-cause mortality | Annualized incidence of mortality during follow-up period until end of data availability; mean follow-up 462 days
  Annualized incidence of all-cause mortality observed from index date (qualifying exacerbation event) through study completion (until end of data availability; mean follow-up 462 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pollack, MS, Study Director — AstraZeneca
Locations (1):
- AstraZeneca, Wilmington, Delaware, United States

REFERENCES:
- See also: D5980R00095 Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5980R00095&attachmentIdentifier=051d686c-8144-48a7-af4a-0e97ee725422&fileName=D5980R00095_Redacted_CSR_Synopsis.pdf&versionIdentifier=